CLINICAL TRIAL: NCT05879757
Title: A Prospective, Observational Study to Assess the Real-World Usage and Outcomes of HyQvia in Patients With Multiple Myeloma (MM) Diagnosed With Secondary Immunodeficiency (SID)
Brief Title: Real-world Usage of HyQvia in Multiple Myeloma Adults With Secondary Immunodeficiency
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-771-5006
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma; Secondary Immunodeficiency (SID)
Keywords: Drug Therapy; Supportive Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MM Participants With SID: Participants with MM diagnosed with SID will be treated with HyQvia as part of routine clinical care and will be followed prospectively from the date of starting HyQvia treatment through 12 months of follow-up.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered in this study.

SUMMARY:
In this study, multiple myeloma participants with secondary immunodeficiency (SID) will be treated with HyQvia according to their clinic's standard practice. The study's main aim is to look into infusion parameters of HyQvia administration.

DETAILED DESCRIPTION:
This is a prospective, observational study of adults having multiple myeloma (MM) with SID treated with HyQvia as part of routine clinical care. This study will characterize the real-world infusion parameters of HyQvia administration.

The study will enroll approximately 100 participants.

Study data will be requested through participants' routine clinic visits and patient-reported outcome (PRO)s are voluntary.

This multi-center trial will be conducted in selected European and South American countries. The overall time of this study is 38 months. Participants will make multiple visits to the clinic within 12 months after enrolment for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria assessed at the time of enrollment are eligible for this study:

1. Ability and willingness to provide informed consent. For adult participants unable to provide informed consent, informed consent provided by the legally authorized representative (LAR).
2. Has a diagnosis of MM requiring systemic anti-myeloma therapy as per International Myeloma Working Group (IMWG) criteria.
3. Initiated HyQvia treatment as part of routine clinical care no more than 30 days before study enrollment or received no more than 2 doses of HyQvia treatment, whichever occurs first. Participants are also eligible if they newly start HyQvia within 30 days after the enrollment visit.

   Note: Participants who do not start HyQvia treatment within 30 days of enrollment will be considered as screen failures (and replaced).
4. Age >=18 years old at the time of MM diagnosis.
5. Available medical history records starting from the diagnosis of MM requiring systemic anti-myeloma therapy as IMWG criteria.
6. Life expectancy >6 months at the time of enrollment, per physician assessment.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of <=2.
8. Participants/LAR willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

Participants who meet any of the following criteria assessed at the time of enrollment are not eligible for this study:

1. Known hypersensitivity to any of the components of HyQvia.
2. Primary immunodeficiency (PID) or diagnosed with human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS) and/or active hepatitis C and/or active hepatitis B infection.
3. Prior use of Ig treatment or prophylaxis within 3 months from the date of enrollment.
4. Serious infection(s) requiring intravenous (IV) treatment at the time of enrollment into the study; except for participants on short-term oral antibiotic therapy.
5. Has participated in an interventional clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in an interventional clinical study involving a medical product or device during this study.

   Note: Participants on investigational chimeric antigen receptor-T (CAR-T) cell therapies and/or bispecific antibodies may participate.
6. Planned stem cell transplant during the treatment period or had a prior stem cell transplant: allogeneic transplant at any time, autologous transplant within 3 months of enrollment.
7. History of malignancy (other than MM) within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, localized prostate cancer or other non-invasive lesion that in the opinion of the investigator, is considered cured with minimal risk of recurrence within 3 years).
8. Participant has had major surgery within 2 weeks before enrollment, or has not fully recovered from an earlier surgery, or has surgery planned during the time the participant is expected to participate in the study.

Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult participants who suffer from MM, have a diagnosis of SID defined according to the European HyQvia label.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2027-02-16 (Estimated); Study Completion 2027-02-16 (Estimated)

PRIMARY OUTCOMES:
Dose of HyQvia per Kilogram of Body Weight | Up to 12 months
  Dose of HyQvia will be calculated as grams per kilogram (g/kg) body weight per 4 weeks.
Absolute Dose of HyQvia per Infusion | Up to 12 months
  Absolute dose of HyQvia will be calculated as dose per infusion in milligrams (mg).
Treatment Interval | Up to 12 months
  Treatment interval and ramp up dosing intervals will be reported as Weekly, every 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks and other administration according to the schedule defined by physician.
Infusion Volume per Site | Up to 12 months
Total Infusion Volume | Up to 12 months
Infusion Rate | Up to 12 months
  Infusion rate will be reported in milliliters per hour (mL/h).
Duration of Infusion | Up to 12 months
  The duration between start and end of infusion will be reported.
Location of Infusion Sites | Up to 12 months
  Location of infusion sites will include right upper abdomen, left upper abdomen, right lower abdomen, left lower abdomen, right or left thigh, right or left arm, and other (specified).
Number of Infusion Sites | Up to 12 months
Number of Participants Characterized by Site of Care | Up to 12 months
  Site of care will be categorized as home, hospital, doctor's office, other (specified).
Length and Diameter of Infusion Needles | Up to 12 months
Number of Participants per Type of Pump | Up to 12 months
  Type of pump will include peristaltic infusion pump and syringe driver pump.
Number of Participants With Availability of Caregiver Support | Up to 12 months
  Availability of caregiver support will be collected as yes, no, and unknown. If yes, caregiver relationship will be specified.
Number of Training Visits | Up to 12 months
Number of Participants With Infusions That are Discontinued, Slowed, or Interrupted | Up to 12 months
Number of Participants With Reasons of infusions Discontinued, Slowed, or Interrupted | Up to 12 months
Number of Participants With Reasons for Discontinued, or Interrupted HyQvia Treatment or Switches to Other Treatment | Up to 12 months
  Reasons for discontinued, or interrupted HyQvia treatment will include local adverse events (AE)/discomfort, systemic AE, administration complexity, insurance/reimbursement-related, low immunoglobulin (Ig) trough level, lack of effectiveness, inability to tolerate large volumes, death and other (specified). If switch, type of treatment after switch (example, antibiotic treatment, intravenous immunoglobulin [IVIg], subcutaneous immunoglobulin [SCIg], unknown) or switches to other treatment will be included.

SECONDARY OUTCOMES:
Time of Multiple Myeloma (MM) Diagnosis | At the time of baseline
Number of Participants Characterized by Clinical Characteristics | Up to 12 months
  Clinical characteristics of participants will include type of MM, and MM treatment/procedures, comorbidities, concomitant medications, laboratory tests and imaging.
Number of Participants Characterized With Type of Hemato-oncological Treatment | Baseline up to 12 months
  Type of hemato-oncological treatment will list type, switches, interruptions and discontinuation with reasons of hemato-oncological treatment or procedure.
Duration of Hemato-oncological Treatment | Baseline up to 12 months
Number of Participants With Multiple Myeloma (MM) Disease Status and Outcome at 12 Months | Month 12
  MM disease status and outcome will include response and criteria used to assess response (if known).
Overall Survival (OS) | Up to 12 months
  OS will be summarized as the frequency and percentage of participants surviving to each follow-up visit. Additionally, time-to death, defined as the time from HyQvia initiation to death occurring before the end of the study period, will be assessed.
Number of Participants With Healthcare Resource Utilization (HCRU) | Up to 12 months
  Number of participants with HCRU including annualized rates and emergency room visits, urgent care visits, outpatient visits, telemedicine visits, and other physician visits, with stratification of hospitalizations and visits due to infection, visit type and provider type.
Duration of Hospitalizations | Up to 12 months
Number of Participants With Related and Not Related Serious Adverse Events (SAEs) | Up to 12 months
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as an untoward medical occurrence that at any dose is fatal, life-threatening, requires inpatient hospitalisation or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event. AEs will be reported as local or systemic AEs.
Number of Participants With Non-serious Adverse Events (AEs) Causally or Temporally Related to HyQvia Treatment | Up to 12 months
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. AEs will be reported as local or systemic AEs.
Number of Participants With Premedication use for HyQvia Infusions, any Technical Problems With the Infusion, and the Planned Versus Actual Dosing | Up to 12 months
  Premedication use for HyQvia infusions will include start date, stop date and medication name. Technical problems with infusion will include problems with the handling of the pump, problems with the preparation of the infusion, problems with the infusion itself, infusion site leakage, and other (specified).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- Instituto Privado de Investigaciones Clinicas de Cordoba, Córdoba, Argentina
- Czechia (2):
  - Fakultni nemocnice Plzen, Pilsen
  - Vseobecna fakultni Nemocnice, Prague
- France (5):
  - CHU Amiens - Hopital Sud, Salouël, Somme
  - CHU Dijon - Hopital du Bocage, Dijon
  - Hopital Prive du Confluent, Nantes
  - Hopital de la Source - CHR Orleans, Orléans
  - CHU Bordeaux - Hopital Haut-Leveque, Pessac
- MHP-Muenchner Haematologiepraxis, Berlin, Germany
- Greece (2):
  - Alexandra General Hospital, Athens
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Italy (4):
  - A.O.U.C Policlinico di Bari, Bari
  - AOU Policlinico Rodolico San Marco, Catania
  - Azienda Ospedale Universita Padova, Padua
  - University of Padova, Treviso
- Pomorski Uniwersytet Medyczny, Szczecin, Poland
- Romania (4):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari Son Espases, Palma
- Lund University Hospital, Lund, Sweden
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Istanbul Universitesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/7f0fdc7891764dc5?idFilter=%5B%22TAK-771-5006%22%5D